CLINICAL TRIAL: NCT03555253
Title: A Pilot Single-Center Study of a Manualized Resilience-Based Telehealth Program for Support Partners of Persons With Multiple Sclerosis
Brief Title: Resilience-Based Program for Support Partners of Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healios Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Halstead, Principal Investigator, Healios Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocol R-PILO-MSOO-010-0002
Record Dates: First submitted 2018-05-14; First posted 2018-06-13 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Resilience; Telehealth; Well-being; Support; Caregiving
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PwMS and their Support Partner (Experimental): Support Partners will participate in six resilience coaching Program Sessions conducted weekly by a study resilience coach. PwMS will participate in the initial and final coaching Program Sessions with their Support Partners.
  Interventions: Behavioral: Resilience-Based Program for Support Partners of PwMS

INTERVENTIONS:
Behavioral: Resilience-Based Program for Support Partners of PwMS — Support Partners will participate in six resilience coaching Program Sessions conducted weekly by a study resilience coach. PwMS will participate in the initial and final coaching Program Sessions with their Support Partners. The MyHealios Resilience Program for PwMS and their Support Partners has been designed to be interactive and include skills-based activities led by the Resilience coach. This includes skills of communication, problem solving, and learning about resilience and cognition in MS.

SUMMARY:
This is a pilot feasibility study to examine the impact of providing a non-therapeutic resilience-based coaching telehealth program to the Support Partners (SP) of persons with MS (PwMS).

Cognitive difficulties are a prominent feature in PwMS and prove to be a challenge for PwMS and the close family members that care for them. This study is a pilot telehealth program that aims to address these needs and improve the overall well-being of adults with MS and their Support Partners.

A manualized program was developed utilizing the previous research study conducted literature, and the expertise and experience of the research study team. Funding was sought and obtained for 30 pairs to participate in the pilot. The 6-session program will address needs identified by this population and improve knowledge of cognition in PwMS.

Study Objectives:

Primary Objective:

To conduct an evaluation of the feasibility of the resilience program by examining:

1. Recruitment (i.e. willingness to participate in program)
2. Participation rates and attrition
3. Participant satisfaction of the program.

Secondary Objective (Support Partner):

To assess the potential long-term benefits of the program to Support Partners of PwMS. Program benefits will be assessed using the following outcomes:

1. Sense of Competencies
2. Understanding of cognitive impairment in MS
3. Caregiver burden
4. Positive Emotions.

Secondary Objective (PwMS):

To assess the potential long-term benefits of the program to PwMS. Program benefits will be assessed using the following outcomes:

1. Relationship Satisfaction
2. Perceived Support.

ELIGIBILITY:
Support Partner Inclusion Criteria

In order to be eligible to participate in this study as a Support Partner, an individual must meet all of the following criteria:

1. Provide signed and dated informed consent form.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Male or female, aged 21 to 65 years.
4. Able to speak, read, and understand English.
5. Reside in the U.S.
6. Live with PwMS who is willing to participate in the study and who meets all of the eligibility criteria.
7. Has access to a telephone and computer or tablet with a stable internet connection as well as a web camera in a private setting.
8. Provide identification that meets the New Jersey Telemedicine Act of 2017.
9. Demonstrate basic ability to use a computer by completing the electronic ICF completion process, which requires use of a teleconferencing platform similar to what will be used during the intervention.

Support Partner Exclusion Criteria

A Support Partner who meets any of the following criteria will be excluded from participation in this study:

1. Professional healthcare worker (e.g., physician, psychologist, social worker, case manager, nurse, home healthcare aide).
2. Dementia, including Alzheimer's and Lewy Bodies Dementia, as screened by CORE Therapy Assessment Form v.2.
3. Reports that PwMS partner is diagnosed with dementia, including Alzheimer's and Lewy Bodies Dementia.
4. Self-report of any change in medication treating bipolar disorder and any psychiatric condition, including a change in dosage, in the previous 6 months and as screened by CORE Therapy Assessment Form v.2.
5. Current suicidal intent as screened by CORE-OM and CORE Therapy Assessment Form v.2.
6. Currently participating in couple or family therapy.
7. An intellectual or developmental disability as screened by CORE Therapy Assessment Form v.2.
8. Evidence of significant brain injury or medical condition leading to cognitive impairment (e.g. accident, tumor) as screened by CORE Therapy Assessment Form v.2.
9. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

PwMS Inclusion Criteria

In order to be eligible to participate in this study as a Person with MS, an individual must meet all of the following criteria:

1. Provide signed and dated informed consent form.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Male or female, aged 21 to 65 years.
4. Self-report of Multiple Sclerosis including the date of the diagnosis (month and year) and the name of the diagnosing physician.
5. Able to speak, read, and understand English.
6. Reside in the U.S.
7. Cognitive difficulty as screened by the PDQ Cognitive Function (score greater than 20).
8. Live with Support Partner who meets all study eligibility criteria.
9. Has access to a telephone and computer or tablet with a stable internet connection as well as a web camera in a private setting.
10. Provide identification that meets the New Jersey Telemedicine Act of 2017.
11. Demonstrate basic ability to use a computer by completing the electronic ICF completion process, which requires use of a teleconferencing platform similar to what will be used during the intervention.

PwMS Exclusion Criteria

A PwMS who meets any of the following criteria will be excluded from participation in this study:

1. Dementia, including Alzheimer's and Lewy Bodies Dementia, as screened by CORE Therapy Assessment Form v.2.
2. Self-report of any change in medication treating bipolar disorder and any psychiatric condition, including a change in dosage, in the previous 6 months and as screened by CORE Therapy Assessment Form v.2.
3. Current suicidal intent as screened by CORE-OM and CORE Therapy Assessment Form v.2.
4. Currently participating in couple or family therapy.
5. Diagnosis of intellectual or developmental disability as screened by CORE Therapy Assessment Form v.2.
6. Significant brain injury or medical condition leading to cognitive impairment (e.g. accident, tumor) as screened by CORE Therapy Assessment Form v.2.
7. Self-report of any change in medication treating MS, including a change dosage, in the previous 3 months.
8. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment (i.e. willingness to participate in program) | Up to 1 year
  Recruitment will end when 30 fully evaluable Support Partner - PwMS pairs have completed the study. It is expected that approximately 45 pairs will be enrolled in order to produce the 30 fully evaluable pairs.
Feasibility: Participation rates and attrition | Up to 1 year
  Participation rates will be measured in terms of individual sessions completed. Attrition rates will be measured. Attrition or drop-out will be addressed as follows: those who drop out prior to the fourth session will be asked to complete a satisfaction questionnaire while those who drop out after the fourth session will be asked to complete post-measures and a satisfaction questionnaire.
Feasibility: Participant satisfaction of the program. | Up to 1 year
  The Intervention Evaluation Questionnaire was created by the research lead as a self-report measure of the participant's evaluation of the intervention and the individual sessions. Participants' evaluation data will be presented as totals from one five-point Likert scale, three yes/no questions and four open questions. The scale question measures satisfaction with the program on a range from 0 (not at all satisfied) to 4 (very satisfied). In addition to this evaluation of the intervention, four questions will be asked at the end of each session to the participants of that session. This includes two five-point Likert scale questions and two open ended questions. The first scale question measures satisfaction with the session on a range from 1 (not at all satisfied) to 5 (very satisfied). The second scale question measures the perceived helpfulness of the session on a range from 1 (not at all satisfied) to 5 (very satisfied).

SECONDARY OUTCOMES:
Change from Baseline: Sense of Competence Questionnaire (Support Partner) | Up to 8 months from enrollment
  The Sense of Competence Questionnaire will be used to measure the support partner's sense of competence in caring for a person with MS. The measure has twenty-seven items. Each item is a statement which the support partner is asked to endorse using a 5-point scale. Response options range from 1 (Yes, completely agrees) to 5 (no, completely disagrees). The three subscales are: satisfaction with care recipient (7 items), satisfaction with one's performance as a support partner (12 items), and consequences of involvement in care for the personal life of the support partner (8 items).
Change from Baseline: Connor-Davidson Resilience Scale (Support Partner) | Up to 8 months from enrollment
  The 10-item version of the Connor-Davidson Resilience Scale will be used to measure the Support Partner's sense of their resilience when faced with stressful situations and negative emotions. The measure includes a total of ten items. Each item on the scale is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Not True at All) to 4 (True Nearly All the Time).
Change from Baseline: Zarit Burden Interview (Support Partner) | Up to 8 months from enrollment
  The Zarit Burden Interview will be used to measure the Support Partner's feelings of burden related to caregiving. There are twenty-two items total. Each item is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).
Change from Baseline: Perceived Stress (Support Partner) | Up to 8 months from enrollment
  The Perceived Stress Survey (PSS) will be used to measure the support partner's perceptions about the nature of events and their relationship to the support partner's values and perceived coping resources. The PSS has 14 items total. Each item is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Very often).
Change from Baseline: Knowledge Questionnaire (Support Partner) | Up to 8 months from enrollment
  The knowledge questionnaire was created by the research lead as a self-report measure of participant retention of the program's topics. The questionnaire has thirteen questions, nine which are multiple-choice questions whose response options are based on the session contents. There are also four scale questions. The first scale question measures the participant's self-reported resilience from 1 (not resilient at all) to 10 (very resilient). The second scale question measures the participant's comfort with their knowledge about cognition in multiple sclerosis from 1 (not comfortable at all) to 10 (very comfortable). The third scale question measures the participant's effectiveness at communicating with their partner from 1 (not effective at all) to 10 (very effective). The fourth scale question measures the participant's effectiveness when using problem-solving skills in dealing with day-to-day difficulties from 1 (not effective at all) to 10 (very effective).
Change from Baseline: Positive and Negative Affect Schedule (Support Partner) | Up to 8 months from enrollment
  The Positive and Negative Affect Schedule will be used to measure the support partner's self-reported experience of positive and negative affect in the past week. The full PANAS has 20 items total. Each item describes an emotion, the recent experience of which (currently at the time of reporting or within the past week) the support partner is asked to endorse using a 5-point scale. Response options range from 1 (feeling the emotion slightly or not at all) or 5 (feeling the emotion often). Ten items describe positive emotion and ten items describe negative emotion.
Change from Baseline: Burns Relationship Satisfaction Scale (Support Partner) | Up to 8 months from enrollment
  The Burns Relationship Satisfaction Scale (BRSS) will be used to assess the support partner's self-reported level of satisfaction in various areas of the relationship with the care recipient for spousal dyads. The BRSS has seven items. Each item describes a relationship area: communication and openness, conflict resolution, degree of caring and affection, intimacy and closeness, satisfaction with roles in relationship, and overall relationship satisfaction. The support partner is asked to rate their degree of satisfaction in each of these areas. Response options range from 0 (very dissatisfied) to 6 (very satisfied).
Change from Baseline: Relationship Assessment Scale (Support Partner) | Up to 8 months from enrollment
  The Relationship Assessment Scale (RAS) will be used to assess the support partner's self-reported level of satisfaction with their relationship with the care recipient. The RAS will only be used in the case of non-spousal dyads. The RAS has seven items. Each item is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 1 (low) to 5 (high). Items 4 and 7 are reverse-scored. Scoring is kept continuous; the higher the score, the more satisfied the respondent is with his/her relationship.
Change from Baseline: Modified Social Support Survey (Person with Multiple Sclerosis) | Up to 8 months from enrollment
  The Modified Social Support Survey (MSSS) will be used to measure the MS participant's perceived social support. The MSSS consists of 18 items. Each item presents a statement that the MS participant is asked to endorse on a 5-point scale. Response options range from 1 (none of the time) to 5 (all of the time). The MSSS has four subscales that measure different dimensions of social support, including tangible support (4 items), emotional support (8 items), affective support (3 items) and positive support (3 items).
Change from Baseline: Burns Relationship Satisfaction Scale (Person with Multiple Sclerosis) | Up to 8 months from enrollment
  The Burns Relationship Satisfaction Scale will be used to assess the MS participant's self-reported level of satisfaction in various areas of the relationship with the support partner for spousal dyads. The BRSS has seven items. Each item describes a relationship area: communication and openness, conflict resolution, degree of caring and affection, intimacy and closeness, satisfaction with roles in relationship, and overall relationship satisfaction. The MS participant is asked to rate their degree of satisfaction in each of these areas. Response options range from 0 (very dissatisfied) to 6 (very satisfied).
Change from Baseline: Relationship Assessment Scale (Person with Multiple Sclerosis) | Up to 8 months from enrollment
  The Relationship Assessment Scale will be used to assess the MS participant's self-reported level of satisfaction with their relationship with the support partner. The RAS will only be used in the case of non-spousal dyads. The RAS has seven items. Each item is a statement which the MS participant is asked to endorse using a 5-point scale. Response options range from 1 (low) to 5 (high). Items 4 and 7 are reverse-scored. Scoring is kept continuous; the higher the score, the more satisfied the respondent is with his/her relationship.

CONTACTS AND LOCATIONS:
Locations (1):
- Healios, Inc., Flemington, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Halstead EJ, Leavitt VM, Fiore D, Mueser KT. A feasibility study of a manualized resilience-based telehealth program for persons with multiple sclerosis and their support partners. Mult Scler J Exp Transl Clin. 2020 Aug 21;6(3):2055217320941250. doi: 10.1177/2055217320941250. eCollection 2020 Jul-Sep. PMID 32913660